CLINICAL TRIAL: NCT03109093
Title: A Multicenter, Single-arm Study to Assess the Efficacy, Safety, and Tolerability of the BiTE® Antibody Blinatumomab in Adult Patients With Minimal Residual Disease (MRD) of B-precursor Acute Lymphoblastic Leukemia (Blast Successor Trial)
Brief Title: Blinatumomab in Adult Patients With Minimal Residual Disease (MRD) of B-precursor Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Principal Investigator, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL-MOLACT1-BLINA; 2015-000733-76 (EudraCT Number)
Record Dates: First submitted 2017-03-13; First posted 2017-04-12 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: ALL, Recurrent, Adult
Keywords: ALL; acute lymphoblastic leukemia; MRD positive; minimal residual disease; blinatumomab
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blinatumomab (Experimental): Patients will receive four cycles of treatment, unless criteria for treatment discontinuation apply. The duration of one cycle is 6 weeks, including a four week continuous intravenous infusion and a two week infusion free interval, which may be extended by a maximum of 7 days.
  Patients entered with MRD level <10-4 (non quantifiable/MolNE1, quantifiable/MolNE2) or positive MRD, non quantifiable (MolNE3) will receive up to two cycles of Blinatumomab.
  Transfer of patients to alloHSCT after one cycle or after subsequent cycles is considered as per protocol discontinuation and as premature treatment discontinuation In case of hematological or extramedullary relapse, the study treatment will be permanently discontinued.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Patients will receive blinatumomab at a dose of 28 µg/day as continuous intravenous infusion at constant flow rate for four weeks, followed by a two-week infusion free interval, defined as one treatment cycle. Up to of four cycles will be performed.
  In case of defined toxicities, the dose of blinatumomab may be reduced to 9µg/day.
  Patients with an MRD relapse may qualify to receive additional treatment with blinatumomab.
  Other Names: blincyto

SUMMARY:
This study is designed to confirm the efficacy, safety, and tolerability of blinatumomab in patients with MRD of B- precursor ALL in complete hematological remission including patients with relapse after SCT. The study aims to expand experience generated in previous trials in patients with MRD positive ALL with a focus on additional specific questions.

DETAILED DESCRIPTION:
Transfer of patients to alloHSCT after one cycle or after a subsequent cycle is considered as per protocol discontinuation and as premature treatment discontinuation.

In case of hematological or extramedullary relapse, the study treatment will be permanently discontinued.

There will be a safety follow-up visit at 30 days after end of the last infusion. There will be efficacy follow-up until 18 months after treatment start. In patients scheduled for SCT the 30-day safety-visit may be performed at the latest time point possible before initiation of subsequent treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD19 positive B-precursor ALL in complete hematological remission defined as less than 5% blasts in bone marrow after at least three intense chemotherapy blocks (e.g., GMALL induction I-II/consolidation I).
2. Presence of minimal residual disease (MRD) after an interval of at least 8 days from last systemic chemo-therapy

   * at a level of ≥10-4 - <10-3 (molecular failure or molecular relapse) in an assay with a minimum sensitivity of 10-4 documented after an interval of at least 2 weeks from last systemic chemotherapy OR
   * at levels below 10-4 documented after an interval of at least 2 weeks from last systemic chemotherapy:

     * Positive <10-4, non quantifiable (MolNE1) OR
     * Positive <10-4 (MolNE2) OR
   * Presence of minimal residual disease (MRD), non quantifiable (MolNE3).
3. For evaluation of MRD patients must have at least one molecular marker based on individual rearrangements of immunoglobulin, TCR-genes or other suitable genes evaluated by the reference laboratory of the trial
4. Bone marrow function as defined below:

   * ANC (Neutrophils) >= 1,000/µL
   * Platelets >= 50,000/µL (transfusion permitted)
   * HB level >= 9g/dl (transfusion permitted)
5. Renal and hepatic function as defined below:

   * AST (GOT), ALT (GPT), and AP < 5 x upper limit of normal (ULN)
   * Total bilirubin < 1.5 x ULN (unless related to Gilbert's Meulengracht disease)
   * Creatinine < 1.5x ULN
   * Creatinine clearance >= 60 mL/min (e.g. calculated according Cockroft&Gault)
6. Negative HIV test, negative hepatitis B (HbsAg) and hepatitis C virus (anti-HCV) test
7. Negative pregnancy test in women of childbearing potential
8. ECOG Performance Status 0 or 1
9. Age >=18 years
10. Ability to understand and willingness to sign a written informed consent
11. Signed and dated written informed consent is available
12. Participation in the registry of the German Multicenter Study Group for Adult ALL (GMALL)

Exclusion Criteria:

1. Ph/BCR-ABL positive ALL
2. Presence of circulating blasts or current extramedullary involvement by ALL
3. History or presence of clinically relevant CNS pathology (e.g. seizure, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome or psychosis)
4. Current detection of ALL blast cells in cerebro-spinal fluid
5. History of or active relevant autoimmune disease
6. Systemic cancer chemotherapy within 2 weeks prior to study treatment (except for intrathecal prophylaxis)
7. Radiotherapy within 4 weeks prior to study treatment
8. Live vaccination within 2 weeks before the start of study treatment
9. Autologous hematopoietic stem cell transplantation (SCT) within six weeks prior to study treatment
10. Allogeneic SCT within 12 weeks before the start of study treatment
11. Any active acute Graft-versus-Host Disease (GvHD), grade 2-4 according to the Glucksberg criteria or active chronic GvHD requiring systemic treatment
12. Any systemic therapy against GvHD within 2 weeks before start of study treatment
13. Therapy with monoclonal antibodies (rituximab, alemtuzumab) within 4 weeks prior to study treatment
14. Treatment with any investigational product within four weeks prior to study treatment
15. Previous treatment with blinatumomab or other anti-CD19-therapy
16. Known hypersensitivity to immunoglobulins or to any other component of the study drug formulation
17. History of malignancy other than ALL diagnosed within 5 years prior to start of protocol-specified therapy with the exception of:

    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated cervical carcinoma in situ without evidence of disease
    * Adequately treated breast ductal carcinoma in situ without evidence of disease
    * Prostatic intraepithelial neoplasia without evidence of prostate cancer
18. Active infection, any other concurrent disease or medical condition that are deemed to interfere with the conduct of the study as judged by the investigator
19. Nursing women
20. Woman of childbearing potential and is not willing to use 2 highly effective methods of contraception while receiving study treatment and for an additional 3 months after the last dose of study treatment.
21. Male who has a female partner of childbearing potential, and is not willing to use 2 highly effective forms of contraception while receiving study treatment and for at least an additional 3 months after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
MRD response after one cycle | after one cycle of treatment (up to 43 days)
  Proportion of patients who achieve complete MRD response after one cycle of treatment with blinatumomab in patients with and without prior SCT

SECONDARY OUTCOMES:
Continuous complete remission | 18 months following initiation of blinatumomab
  Probability of continuous complete remission (remission duration) at 18 months following initiation of blinatumomab (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
Hematological relapse-free survival | 18 months following initiation of blinatumomab
  Probability of hematological relapse-free survival rate at 18 months following initiation of blinatumomab (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
Overall survival | 18 months following initiation of blinatumomab
  Probability of overall survival at 18 months following initiation of blinatumomab (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
Relapse localisations | In Case of Relapse, continuously until End of Follow-Up (up to 18 Months)
  Frequency of different relapse localisations in proportion to total hematological relapses (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
Biological evaluation of hematological and extramedullary relapse | In Case of Relapse, continuously until End of Follow-Up (up to 18 Months)
  Biological evaluation of hematological and extramedullary relapses including CD19 expression (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
Serious Adverse Event (SAE) incidence | continuously until End of Safety-Follow-Up (up to 26 weeks)
  Overall incidence and severity of adverse events in patients with and without prior SCT (CTCAE 4.0) (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
MRD response after two cycles | after two cycles of treatment (up to 85 days)
  Proportion of patients who achieve MRD response after one or two cycles of treatment with Blinatumomab (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
complete MRD response after two cycles | after two cycles of treatment (up to 85 days)
  Proportion of patients who achieve complete MRD response after two cycles of treatment with blinatumomab in patients with and without prior SCT (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
duration of MRD response | 18 months following initiation of blinatumomab
  Probability of continuous MRD response and complete MRD response and duration of MRD response at 18 months following initiation of blinatumomab (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
Time to MRD response | MRD determination after each cycle of treatment (up to 24 weeks)
  Time to MRD response measured by time-point of first achievement (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
GvHD | until End of Safety-Follow-Up (up to 26 weeks)
  Evaluation of GvHD as part of AE documentation and according to Glucksberg Criteria, grade and localisation. (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
treatment related mortality after subsequent SCT | after subsequent SCT (at day 100 and later)
  Evaluation of overall survival, remission duration, relapse-free survival and treatment related mortality (at day 100 and later) in patients with SCT in complete remission after blinatumomab (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
treatment related mortality | continuously until End of Follow-Up (up to 18 Months)
  Evaluation of overall survival, remission duration, relapse-free survival and treatment related mortality in patients without SCT in complete remission after blinatumomab (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)
Quality of Life | until End of Follow-Up (up to 18 Months)
  Measurement of Quality of Life with EORTC instruments (EORTC QLQ C30 and EQ-5D) at different time-points during treatment (Separate analysis of all outcome parameters in patients with MRD above 10-4, 10-4-10-3 and patients with MRD below 10-4 or non-quantifiable MRD)

OTHER OUTCOMES:
Treatment deviation1 | until end of treatment (up to 22 weeks)
  Incidence of dose reductions
Treatment deviation2 | until end of treatment (up to 22 weeks)
  incidence of treatment interruptions
Treatment deviation3 | until end of treatment (up to 22 weeks)
  days of interruption
Treatment deviation4 | until end of treatment (up to 22 weeks)
  withdrawals
Treatment deviation5 | until end of treatment (up to 22 weeks)
  total delivered dose
Treatment deviation6 | until end of treatment (up to 22 weeks)
  total days of treatment
Treatment deviation7 | until end of treatment (up to 22 weeks)
  realisation rate calculated as scheduled total dose/delivered total dose
Hospitalisation days | until end of treatment (up to 22 weeks)
  Number of hospitalisation days

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Goekbuget, MD, Principal Investigator — GMALL-Study-Group
Locations (22):
- Germany (22):
  - University Hospital of Frankfurt (Main), Frankfurt am Main, Hesse
  - Charité - Campus Benjamin Franklin, Berlin
  - Uniklinik Dresden, Dresden
  - Uniklinik Düsseldorf, Düsseldorf
  - Univeristätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Uniklinik Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Uniklinik Heidelberg, Heidelberg
  - UKSH-Kiel, Kiel
  - Universitätsklinik Leipzig, Leipzig
  - Klinikum Mannheim, Mannheim
  - Universitätsklinkum Gießen und Marburg, Marburg
  - Klinikum Großhadern, München
  - Uniklinik Münster, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Uniklinik Regensburg, Regensburg
  - Robert - Bosch - Krankenhaus, Stuttgart
  - Universitätsklinik Tübingen, Tübingen
  - Universitätsklinkum Ulm, Ulm
  - Uniklinik Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gökbuget N, et al . Interim Results of a Multicenter, Single-Arm Study to Assess Blinatumomab in Adult Patients (pts) with Minimal Residual Disease (MRD) of B-Precursor (BCP) Acute Lymphoblastic Leukemia (GMALL-MOLACT1-BLINA). Blood (2020) 136 (Supplement 1): 39-40.